CLINICAL TRIAL: NCT00716937
Title: Recurrence, Complications, Work-off Date, Healing Time and Patients Willingness in Karydakis Technique for Treatment of Sacrococcygeal Pilonidal Sinus Versus Excision With Healing by Secondary Intention (EHSI)Technique
Brief Title: Karydakis Procedure Versus Excision With Healing by Secondary Intention (EHSI) in Sacrococcygeal Pilonidal Sinus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6148; 86-04-30-6148 (Other: Tehran University of Medical Sciences)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Pilonidal Sinus; Pilonidal Cyst
Keywords: pilonidal sinus; karydakis; laying open
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Excision of the cyst and Karydakis flap
  Interventions: Procedure: karydakis flap
- 2 (Experimental): Excision of the cyst and laying open
  Interventions: Procedure: karydakis flap; Procedure: laying open

INTERVENTIONS:
Procedure: karydakis flap — Karydakis flap is a type of primary repair of the wound, after complete excision of sacral pilonidal cyst with 2 characteristics 1)lateralization of final scar 2)flattening of natal cleft
  Other Names: lateralization; primary repair
Procedure: laying open — laying open the site of excision of sinus or cyst without any flap
  Arms: 2

SUMMARY:
Recurrence, Complications, Work-off date, Healing time and Patients Willingness in Karydakis Technique for Treatment of Sacrococcygeal Pilonidal Sinus versus Healing by Secondary Intention (EHSI) Technique in Imam Khomeini Hospital from 2008 to 2011

ELIGIBILITY:
Inclusion Criteria:

all types of pilonidal sinus or cyst

Exclusion Criteria:

no exclusion criteria

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2007-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Recurrence | 1 year after surgery

SECONDARY OUTCOMES:
Work off date, Healing Time | up to 1 Year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amir Keshvari, Assoc. Prof., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of medical Sciences, Deputy of Research, Tehran, Tehran Province, Iran